CLINICAL TRIAL: NCT00661713
Title: A Phase 2b/3, Multi-Center, Observer-Blind, Controlled Study of the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine Administered to Healthy Adolescents Aged 11-17 Years According to Different Vaccination Schedules
Brief Title: Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine Administered to Healthy Adolescents According to Different Vaccination Schedules
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V72P10
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Meningococcal Disease
Keywords: Meningococcal disease; Neisseria meningitidis serogroup B; prevention; vaccination; adolescents
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant

ARMS (8):
- rMenB06 (Experimental): Subjects received one injection of rMenB+OMV NZ vaccine (month 0) and two injections of placebo (at month 1, month 2). A second injection of rMenB+OMV NZ vaccine was given later (month 6).
  Interventions: Biological: rMenB+OMV NZ; Biological: Placebo
- rMenB0 (Experimental): Subjects received one injection of rMenB+OMV NZ vaccine (month 0) and three injections of placebo (month 1, month 2 and month 6).
  Interventions: Biological: rMenB+OMV NZ; Biological: Placebo
- rMenB016 (Experimental): Subjects received two injections of rMenB+OMV NZ vaccine (at month 0 and month 1) and one injection of placebo (at month 2). A third injection of rMenB+OMV NZ vaccine was given later (at month 6).
  Interventions: Biological: rMenB+OMV NZ; Biological: Placebo
- rMenB01 (Experimental): Subjects received two injections of rMenB+OMV NZ vaccine (at month 0 and month 1) and two injection of placebo (at month 2 and month 6).
  Interventions: Biological: rMenB+OMV NZ; Biological: Placebo
- rMenB026 (Experimental): Subjects received two injections of rMenB+OMV NZ vaccine (at month 0 and month 2) and one injection of placebo (at month 2). A third injection of rMenB+OMV NZ vaccine was given later (at month 6).
  Interventions: Biological: rMenB+OMV NZ; Biological: Placebo
- rMenB02 (Experimental): Subjects received two injections of rMenB+OMV NZ vaccine (at month 0 and month 2) and two injections of placebo (at month 1 and month 6).
  Interventions: Biological: rMenB+OMV NZ; Biological: Placebo
- rMenB012 (Experimental): Subjects received three injections of rMenB+OMV NZ vaccine (at month 0, month 1 and month 2) and one injection of placebo later (at month 6).
  Interventions: Biological: rMenB+OMV NZ; Biological: Placebo
- rMenB6 (Experimental): Subjects received three injections of placebo(at month 0, month 1 and month 2) and one injection of rMenB+OMV NZ vaccine(at month 6).
  Interventions: Biological: rMenB+OMV NZ; Biological: Placebo

INTERVENTIONS:
Biological: rMenB+OMV NZ
  Other Names: Serogroup B Meningococcal Vaccine
Biological: Placebo

SUMMARY:
The proposed study is aimed to assess the antibody response and short-term persistence of Novartis Meningococcal B Vaccine after one, two or three doses and to evaluate the optimal vaccination schedule in an adolescent population.

ELIGIBILITY:
Inclusion Criteria:

1)11-17 years of age inclusive who have given their written assent and whose parents or legal guardians have given written informed consent at the time of enrollment;

2)who are available for all the visits scheduled in the study (i.e., not planning to leave the area before the end of the study period);

3)in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. History of any meningococcal B vaccine administration;
2. Current or previous, confirmed or suspected disease caused by N. meningitidis;
3. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrollment;
4. Significant acute or chronic infection within the previous 7 days or fever (defined as axillary temperature ≥38°C) within the previous day;
5. Antibiotics within 6 days prior to enrollment;
6. Pregnancy or nursing (breastfeeding) mothers;
7. Females of childbearing age who have not used or do not plan to use acceptable birth control measures, for the 7 months duration of the study. Oral, injected or implanted hormonal contraceptive, diaphragm, condom, intrauterine device or sexual abstinence are considered acceptable forms of birth control. If sexually active the subject must have been using one of the accepted birth control methods at least two months prior to study entry;
8. Any serious chronic or progressive disease (e.g., neoplasm, diabetes, cardiac disease, hepatic disease, progressive neurological disease or seizure disorder; autoimmune disease, HIV infection or AIDS, or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition).
9. Known or suspected impairment/alteration of the immune system, immunosuppressive therapy, including use of corticosteroids in immunosuppressive doses or chronic use of inhaled high-potency corticosteroids within the previous 60 days. [Use of topical corticosteroids administered during the study in limited areas (i.e., eczema on knees or face or elbows) of the body is allowed]; immunostimulants;
10. Receipt of blood, blood products and/or plasma derivatives, or a parenteral immunoglobulin preparation within the previous 90 days;
11. History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component;
12. Receipt of or intent to immunize with any other vaccine(s) within 30 days prior (60 days for live viral vaccines) and throughout the study period (exception: licensed fluvaccine should not be administered within 14 days prior to enrollment; routine vaccine administration may be administered after the blood draw at Study Month 7);
13. Participation in another clinical trial within the last 90 days or planned for during study;
14. Family members and household members of research staff;
15. Any condition which in the opinion of the investigator and/or the Regional MD may interfere with the evaluation of the study objectives.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1631 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (10):
- Chile (10):
  - Site 13: Liceo Diego Aracena de Lo Barnechea, Monseñor Escrivá de Balaguer 14630, Lo Barnechea, Santiago Metropolitan
  - Site 41: Colegio Antonio Hermida Fabres, Av. Coronel Alejandro Sepúlveda N° 6801
  - Site 43: Liceo José Victorino Lastarria, Av. Miguel Claro N° 32
  - Site 51: Centro Para vacunas en Desarrollo. Hospital de Niños Roberto del Rio, Av. Prof Zañartu 1085
  - Site 15: Liceo Carmela Carvajal de Prat, Avda. Italia 980
  - Site 14: Colegio Parroquial Santa Rosa de Lo Barnechea, Avda. Raúl Labbé Nº 13.799
  - Site 42: Centro Educacional Eduardo de la Barra, Calle A, N° 6301
  - Site 61: Facultad de Medicina. Universidad de Valparaíso., Hontaneda # 2653. Valparaíso
  - Site 11: Complejo Educacional Eduardo Cuevas Valdés, Lo Barnechea
  - Site 12: Colegio San Jose de Lo Barnechea, Santiago

REFERENCES:
- [Derived] Bartolini E, Borgogni E, Bruttini M, Muzzi A, Giuliani M, Iozzi S, Petracca R, Martinelli M, Bonacci S, Marchi S, Brettoni C, Donati C, Torricelli G, Guidotti S, Domina M, Beninati C, Teti G, Felici F, Rappuoli R, Castellino F, Del Giudice G, Masignani V, Pizza M, Maione D. Immunological fingerprint of 4CMenB recombinant antigens via protein microarray reveals key immunosignatures correlating with bactericidal activity. Nat Commun. 2020 Oct 5;11(1):4994. doi: 10.1038/s41467-020-18791-0. PMID 33020485
- [Derived] Santolaya ME, O'Ryan ML, Valenzuela MT, Prado V, Vergara R, Munoz A, Toneatto D, Grana G, Wang H, Clemens R, Dull PM; V72P10 Meningococcal B Adolescent Vaccine Study group. Immunogenicity and tolerability of a multicomponent meningococcal serogroup B (4CMenB) vaccine in healthy adolescents in Chile: a phase 2b/3 randomised, observer-blind, placebo-controlled study. Lancet. 2012 Feb 18;379(9816):617-24. doi: 10.1016/S0140-6736(11)61713-3. Epub 2012 Jan 18. PMID 22260988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 10 study centers in Chile.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- rMenB06: Subjects received 2 doses each of rMenB+OMV-NZ at 0 and 6 months and placebo at 1 and 2 months.
- rMenB0: Subjects received 1 dose of rMenB+OMV-NZ at 0 month and 3 doses of placebo at 1, 2 and 6 months.
- rMenB016: Subjects received 3 doses of rMenB+OMV-NZ at 0, 1 and 6 months and 1 dose of placebo at 2 months.
- rMenB01: Subjects received 2 doses each of rMenB+OMV-NZ at 0 and 1 months and placebo at 2 and 6 months.
- rMenB026: Subjects received 3 doses of rMenB+OMV-NZ at 0, 2 and 6 months and 1 dose of placebo at 1 month.
- rMenB02: Subjects received 2 doses each of rMenB+OMV-NZ at 0 and 2 months and placebo at 1 and 6 months.
- rMenB012: Subjects received 3 doses of rMenB+OMV-NZ at 0, 1 and 2 months and placebo at 6 months.
- rMenB6: Subjects received 1 dose of rMenB+OMV-NZ at 6 months and 3 doses of placebo at 0, 1 and 2 months.
Period: Overall Study
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Started | 128 | 247 | 128 | 247 | 127 | 253 | 373 | 128
Completed | 112 | 208 | 111 | 219 | 107 | 216 | 309 | 117
Not Completed | 16 | 39 | 17 | 28 | 20 | 37 | 64 | 11
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Unable to Classify | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 6 | 3 | 3 | 0 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 11 | 25 | 12 | 21 | 12 | 26 | 45 | 9
Not completed — Lost to Follow-up | 2 | 7 | 2 | 2 | 5 | 7 | 14 | 1
Not completed — Administrative Reason | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Inappropriate Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6 | Total
Number analyzed (Participants) | 128 | 247 | 128 | 247 | 127 | 253 | 373 | 128 | 1631
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.9) | 13.8 (1.9) | 13.9 (1.9) | 13.9 (1.9) | 13.7 (1.9) | 13.7 (1.8) | 13.8 (1.9) | 13.8 (2) | 13.8 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 147 | 76 | 138 | 73 | 138 | 199 | 66 | 913
  Male | 52 | 100 | 52 | 109 | 54 | 115 | 174 | 62 | 718

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With hSBA Titer ≥1:4 After Receiving One, Two or Three Doses of rMenB+OMV NZ Vaccine.
Description: Immunogenicity was evaluated by measuring the percentage of subjects with hSBA titter >1:4 against 44/76-SL, 5/99, NZ98/254 strains at months 1, 2, 3.
Time Frame: Month-1, 2, 3
Population: Analysis was performed as per the protocol dataset
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 334 | 116
percentage of Subjects
  44/76-SL- Mo 0 | 42 [33 to 52] | 47 [40 to 54] | 41 [32 to 50] | 38 [32 to 45] | 37 [28 to 47] | 47 [40 to 53] | 46 [41 to 52] | 46 [36 to 55]
  44/76-SL- Mo 1: number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  44/76-SL- Mo 1 | 92 [85 to 96] | 92 [88 to 95] | 95 [89 to 98] | 93 [88 to 96] | 90 [83 to 95] | 92 [88 to 95] | 95 [92 to 97] | 43 [34 to 53]
  44/76-SL- Mo 2: number analyzed (Participants) | 108 | 213 | 108 | 222 | 105 | 219 | 307 | 109
  44/76-SL- Mo 2 | 88 [80 to 93] | 92 [88 to 95] | 100 [97 to 100] | 100 [98 to 100] | 88 [80 to 93] | 89 [85 to 93] | 100 [98 to 100] | 50 [40 to 59]
  44/76-SL- Mo 3: number analyzed (Participants) | 107 | 208 | 105 | 215 | 104 | 215 | 303 | 108
  44/76-SL- Mo 3 | 84 [76 to 90] | 88 [82 to 92] | 99 [95 to 100] | 100 [97 to 100] | 100 [97 to 100] | 100 [98 to 100] | 100 [98 to 100] | 48 [38 to 58]
  5/99- Mo 0 | 29 [20 to 38] | 41 [35 to 48] | 28 [20 to 38] | 31 [25 to 38] | 30 [22 to 39] | 37 [31 to 44] | 36 [30 to 41] | 29 [21 to 38]
  5/99- Mo 1: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  5/99- Mo 1 | 97 [92 to 99] | 96 [93 to 98] | 96 [90 to 99] | 97 [94 to 99] | 97 [92 to 99] | 95 [92 to 98] | 97 [94 to 98] | 35 [26 to 44]
  5/99- Mo 2: number analyzed (Participants) | 108 | 213 | 108 | 222 | 105 | 219 | 308 | 109
  5/99- Mo 2 | 95 [90 to 98] | 94 [90 to 97] | 100 [97 to 100] | 100 [98 to 100] | 97 [92 to 99] | 96 [93 to 98] | 100 [98 to 100] | 31 [23 to 41]
  5/99- Mo 3: number analyzed (Participants) | 107 | 209 | 105 | 215 | 105 | 215 | 303 | 108
  5/99- Mo 3 | 92 [85 to 96] | 89 [84 to 93] | 99 [95 to 100] | 100 [98 to 100] | 98 [93 to 100] | 100 [98 to 100] | 100 [99 to 100] | 32 [24 to 42]
  NZ98/254-mo 0: number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 333 | 116
  NZ98/254-mo 0 | 32 [24 to 42] | 39 [33 to 46] | 33 [24 to 42] | 35 [29 to 41] | 34 [25 to 43] | 37 [31 to 44] | 33 [28 to 38] | 38 [29 to 47]
  NZ98/254-mo 1: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  NZ98/254-mo 1 | 90 [83 to 95] | 94 [90 to 97] | 95 [89 to 98] | 94 [90 to 96] | 90 [83 to 95] | 93 [89 to 96] | 95 [92 to 97] | 38 [29 to 48]
  NZ98/254-mo 2: number analyzed (Participants) | 107 | 213 | 108 | 222 | 105 | 218 | 308 | 109
  NZ98/254-mo 2 | 81 [73 to 88] | 84 [74 to 88] | 99 [95 to 100] | 100 [98 to 100] | 78 [69 to 86] | 85 [79 to 89] | 100 [98 to 100] | 39 [29 to 48]
  NZ98/254-mo 3: number analyzed (Participants) | 107 | 208 | 105 | 215 | 104 | 215 | 302 | 108
  NZ98/254-mo 3 | 80 [72 to 87] | 76 [70 to 82] | 97 [92 to 99] | 97 [94 to 99] | 100 [97 to 100] | 100 [98 to 100] | 99 [97 to 100] | 43 [33 to 52]

2. Primary Outcome: Number of Subjects With Local Reactions and Systemic Reactions Occurring in Days 1 to 7 After Vaccination
Description: Safety was assessed as the number of subjects who reported local and systemic reactions during day 1 to day 7 after any vaccination with rMenB+OMV
Time Frame: 1 to 7 days after each vaccination
Population: Analysis was performed as per the safety dataset.
Measure: Number; unit: participants
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 128 | 247 | 128 | 247 | 127 | 253 | 373 | 128
participants
  erythema (local) | 93 | 162 | 95 | 188 | 94 | 172 | 282 | 85
  Induration (Local) | 71 | 130 | 75 | 151 | 82 | 121 | 228 | 57
  Swelling (Local) | 72 | 132 | 81 | 144 | 76 | 115 | 226 | 54
  Pain (Local) | 122 | 236 | 124 | 237 | 113 | 236 | 345 | 123
  Med.Att Fever (Systemic) | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 1
  Malaise (Systemic) | 92 | 181 | 96 | 172 | 87 | 185 | 272 | 89
  Myalgia(Systemic) | 85 | 141 | 91 | 156 | 81 | 160 | 238 | 91
  Arthralgia(Systemic) | 55 | 76 | 55 | 80 | 39 | 105 | 146 | 43
  Headache(Systemic) | 79 | 139 | 88 | 160 | 73 | 165 | 244 | 74
  Nausea(Systemic) | 41 | 80 | 51 | 72 | 42 | 88 | 143 | 49
  Fever(Systemic) | 12 | 8 | 11 | 21 | 18 | 26 | 38 | 18

3. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥1:4 After Receiving a Booster Dose of rMenB+OMV NZ Vaccine at Month 6.
Description: Immunogenicity was evaluated by measuring the percentage of subjects with hSBA titter >1:4 agains 44/76-SL, 5/99, NZ98/254 strains at months 6 & 7.
Time Frame: Month-6 & 7
Population: Analysis was performed as per the protocol dataset.
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 100 | 188 | 100 | 198 | 99 | 201 | 278 | 100
percentage of Subjects
  44/76-SL- Mo 6 | 76 [66 to 84] | 72 [65 to 79] | 93 [86 to 97] | 92 [88 to 96] | 97 [91 to 99] | 98 [94 to 99] | 97 [94 to 99] | 46 [36 to 56]
  44/76-SL- Mo 7: number analyzed (Participants) | 86 | 173 | 95 | 186 | 91 | 179 | 255 | 95
  44/76-SL- Mo 7 | 100 [96 to 100] | 71 [64 to 78] | 100 [96 to 100] | 90 [85 to 94] | 100 [96 to 100] | 95 [91 to 98] | 95 [92 to 98] | 93 [85 to 97]
  5/99- Mo 6 | 79 [70 to 87] | 74 [67 to 80] | 99 [95 to 100] | 98 [96 to 100] | 99 [95 to 100] | 100 [97 to 100] | 100 [98 to 100] | 28 [19 to 38]
  5/99- Mo 7: number analyzed (Participants) | 86 | 173 | 95 | 187 | 91 | 179 | 255 | 95
  5/99- Mo 7 | 99 [94 to 100] | 67 [60 to 74] | 100 [96 to 100] | 98 [95 to 99] | 100 [96 to 100] | 99 [96 to 100] | 99 [97 to 100] | 93 [85 to 97]
  NZ98/254-mo 6: number analyzed (Participants) | 99 | 188 | 100 | 198 | 99 | 200 | 278 | 100
  NZ98/254-mo 6 | 81 [72 to 88] | 69 [62 to 76] | 93 [86 to 97] | 89 [84 to 93] | 97 [91 to 99] | 96 [92 to 98] | 97 [94 to 99] | 45 [35 to 55]
  NZ98/254-mo 7: number analyzed (Participants) | 86 | 172 | 95 | 187 | 91 | 179 | 255 | 95
  NZ98/254-mo 7 | 100 [96 to 100] | 67 [60 to 74] | 100 [96 to 100] | 85 [79 to 90] | 100 [96 to 100] | 94 [89 to 97] | 95 [92 to 98] | 93 [85 to 97]

4. Secondary Outcome: Percentage of Subjects With hSBA Titer ≥1:8 After Primary and Booster Vaccination.
Description: Immunogenicity was evaluated by measuring the percentage of subjects with hSBA titer ≥1:8 against 44/76-SL, 5/99, NZ98/254 strains.
Time Frame: at baseline, month-1, month-2, month-3, month-6 and month-7.
Population: Analysis was performed as per the protocol dataset.
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 334 | 116
percentage of Subjects
  44/76-SL- Mo 0 | 29 [21 to 39] | 37 [31 to 44] | 31 [23 to 40] | 32 [26 to 38] | 30 [22 to 39] | 35 [29 to 42] | 33 [28 to 38] | 33 [24 to 42]
  44/76-SL- Mo 1: number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  44/76-SL- Mo 1 | 87 [79 to 92] | 87 [82 to 91] | 85 [77 to 91] | 85 [80 to 89] | 81 [72 to 88] | 87 [82 to 91] | 86 [82 to 90] | 30 [22 to 40]
  44/76-SL- Mo 2: number analyzed (Participants) | 108 | 213 | 108 | 222 | 105 | 219 | 307 | 109
  44/76-SL- Mo 2 | 79 [70 to 86] | 84 [78 to 89] | 99 [95 to 100] | 99 [97 to 100] | 80 [71 to 87] | 80 [74 to 85] | 99 [98 to 100] | 33 [24 to 43]
  44/76-SL- Mo 3: number analyzed (Participants) | 107 | 208 | 105 | 215 | 104 | 215 | 303 | 108
  44/76-SL- Mo 3 | 74 [64 to 82] | 77 [71 to 83] | 99 [95 to 100] | 98 [95 to 99] | 99 [95 to 100] | 100 [98 to 100] | 99 [97 to 100] | 36 [27 to 46]
  44/76-SL- Mo 6: number analyzed (Participants) | 100 | 188 | 100 | 198 | 99 | 201 | 278 | 100
  44/76-SL- Mo 6 | 62 [52 to 72] | 62 [54 to 69] | 90 [82 to 95] | 83 [77 to 88] | 90 [82 to 95] | 91 [86 to 95] | 93 [90 to 96] | 34 [25 to 44]
  44/76-SL- Mo 7: number analyzed (Participants) | 86 | 173 | 95 | 186 | 91 | 179 | 255 | 95
  44/76-SL- Mo 7 | 99 [94 to 100] | 57 [49 to 64] | 100 [96 to 100] | 82 [75 to 87] | 100 [96 to 100] | 88 [82 to 92] | 91 [86 to 94] | 89 [81 to 95]
  5/99- Mo 0 | 18 [11 to 26] | 24 [19 to 30] | 20 [13 to 29] | 22 [17 to 28] | 23 [15 to 32] | 22 [17 to 28] | 22 [17 to 26] | 14 [8 to 21]
  5/99- Mo 1: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  5/99- Mo 1 | 96 [91 to 99] | 91 [87 to 95] | 89 [82 to 94] | 94 [90 to 96] | 91 [84 to 96] | 93 [89 to 96] | 94 [91 to 96] | 19 [12 to 28]
  5/99- Mo 2: number analyzed (Participants) | 108 | 213 | 108 | 222 | 105 | 219 | 308 | 109
  5/99- Mo 2 | 89 [81 to 94] | 85 [80 to 90] | 100 [97 to 100] | 100 [98 to 100] | 78 [69 to 86] | 88 [83 to 92] | 99 [98 to 100] | 17 [11 to 26]
  5/99- Mo 3: number analyzed (Participants) | 107 | 209 | 105 | 215 | 105 | 215 | 303 | 108
  5/99- Mo 3 | 81 [73 to 88] | 77 [71 to 83] | 99 [95 to 100] | 100 [97 to 100] | 98 [93 to 100] | 100 [98 to 100] | 100 [99 to 100] | 19 [12 to 27]
  5/99- Mo 6: number analyzed (Participants) | 100 | 188 | 100 | 198 | 99 | 201 | 278 | 100
  5/99- Mo 6 | 60 [50 to 70] | 57 [50 to 64] | 97 [91 to 99] | 98 [95 to 99] | 98 [93 to 100] | 99 [96 to 100] | 99 [97 to 100] | 16 [9 to 25]
  5/99- Mo 7: number analyzed (Participants) | 86 | 173 | 95 | 187 | 91 | 179 | 255 | 95
  5/99- Mo 7 | 99 [94 to 100] | 48 [40 to 56] | 100 [96 to 100] | 97 [93 to 99] | 100 [96 to 100] | 97 [94 to 99] | 98 [95 to 99] | 86 [78 to 93]
  NZ98/254 Mo 0: number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 333 | 116
  NZ98/254 Mo 0 | 22 [15 to 31] | 30 [24 to 36] | 27 [19 to 36] | 25 [20 to 31] | 24 [16 to 33] | 26 [21 to 32] | 25 [20 to 30] | 29 [21 to 38]
  NZ98/254 Mo 1: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  NZ98/254 Mo 1 | 84 [76 to 90] | 83 [77 to 87] | 82 [74 to 89] | 84 [79 to 88] | 75 [65 to 82] | 80 [74 to 85] | 86 [81 to 89] | 26 [18 to 35]
  NZ98/254 Mo 2: number analyzed (Participants) | 107 | 213 | 108 | 222 | 105 | 218 | 308 | 109
  NZ98/254 Mo 2 | 72 [62 to 80] | 70 [64 to 76] | 98 [93 to 100] | 99 [97 to 100] | 65 [55 to 74] | 75 [68 to 80] | 99 [97 to 100] | 31 [23 to 41]
  NZ98/254 Mo 3: number analyzed (Participants) | 107 | 208 | 105 | 215 | 104 | 215 | 302 | 108
  NZ98/254 Mo 3 | 70 [60 to 79] | 65 [58 to 71] | 90 [82 to 95] | 91 [86 to 94] | 98 [93 to 100] | 100 [97 to 100] | 98 [96 to 99] | 30 [21 to 39]
  NZ98/254 Mo 6: number analyzed (Participants) | 99 | 188 | 100 | 198 | 99 | 200 | 278 | 100
  NZ98/254 Mo 6 | 60 [49 to 69] | 54 [47 to 62] | 80 [71 to 87] | 77 [70 to 82] | 86 [77 to 92] | 86 [80 to 90] | 91 [87 to 94] | 38 [28 to 48]
  NZ98/254 Mo 7: number analyzed (Participants) | 86 | 172 | 95 | 187 | 91 | 179 | 255 | 95
  NZ98/254 Mo 7 | 99 [94 to 100] | 49 [42 to 57] | 99 [94 to 100] | 71 [64 to 78] | 100 [96 to 100] | 81 [74 to 86] | 84 [79 to 88] | 86 [78 to 93]

5. Secondary Outcome: Percentages of Subjects With at Least a Fourfold Rise in hSBA Titer Over the Prevaccination and After Booster Vaccination.
Description: Immunogenicity was evaluated by measuring the percentage of subjects with at least a fourfold rise in hSBA titer over the prevaccination and after booster vaccination against 44/76-SL, 5/99, NZ98/254 strains at month-1, month-2, month-3 and month-7.
Time Frame: Month-1, month-2, month-3 and month-7
Population: Analysis was performed as per the protocol dataset.
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 333 | 115
percentage of Subjects
  44/76-SL Mo 1 | 73 [64 to 81] | 75 [69 to 80] | 71 [61 to 79] | 77 [71 to 82] | 67 [58 to 76] | 73 [67 to 79] | 72 [67 to 77] | 3 [1 to 7]
  44/76-SL Mo 2: number analyzed (Participants) | 108 | 213 | 107 | 222 | 105 | 219 | 307 | 109
  44/76-SL Mo 2 | 62 [52 to 71] | 67 [60 to 73] | 94 [88 to 98] | 96 [92 to 98] | 65 [55 to 74] | 61 [54 to 67] | 94 [91 to 97] | 6 [2 to 12]
  44/76-SL Mo 3: number analyzed (Participants) | 107 | 208 | 104 | 215 | 104 | 215 | 303 | 108
  44/76-SL Mo 3 | 53 [43 to 63] | 59 [52 to 66] | 88 [81 to 94] | 91 [87 to 95] | 91 [84 to 96] | 95 [92 to 98] | 95 [92 to 97] | 3 [1 to 8]
  44/76-SL Mo 7: number analyzed (Participants) | 86 | 173 | 94 | 186 | 91 | 179 | 255 | 95
  44/76-SL Mo 7 | 95 [89 to 99] | 33 [26 to 40] | 98 [93 to 100] | 73 [66 to 79] | 93 [86 to 98] | 76 [69 to 82] | 80 [75 to 85] | 76 [66 to 84]
  5/99 Mo 1: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  5/99 Mo 1 | 87 [80 to 93] | 79 [73 to 84] | 81 [72 to 87] | 85 [80 to 89] | 79 [70 to 86] | 85 [80 to 89] | 85 [80 to 88] | 3 [1 to 7]
  5/99 Mo 2: number analyzed (Participants) | 108 | 213 | 107 | 222 | 105 | 219 | 308 | 109
  5/99 Mo 2 | 78 [69 to 85] | 65 [58 to 72] | 98 [93 to 100] | 98 [95 to 100] | 63 [53 to 72] | 74 [68 to 80] | 98 [96 to 99] | 5 [2 to 10]
  5/99 Mo 3: number analyzed (Participants) | 107 | 209 | 104 | 215 | 105 | 215 | 303 | 108
  5/99 Mo 3 | 65 [56 to 74] | 53 [46 to 60] | 95 [89 to 98] | 99 [96 to 100] | 96 [91 to 99] | 99 [96 to 100] | 99 [98 to 100] | 6 [3 to 13]
  5/99- Mo 7: number analyzed (Participants) | 86 | 173 | 94 | 187 | 91 | 179 | 255 | 95
  5/99- Mo 7 | 98 [92 to 100] | 27 [21 to 34] | 99 [94 to 100] | 88 [82 to 92] | 99 [94 to 100] | 90 [85 to 94] | 94 [90 to 97] | 82 [73 to 89]
  NZ98/254 Mo 1: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 332 | 115
  NZ98/254 Mo 1 | 72 [63 to 80] | 70 [63 to 76] | 65 [56 to 74] | 74 [67 to 79] | 59 [49 to 68] | 64 [58 to 70] | 73 [68 to 78] | 3 [1 to 7]
  NZ98/254 Mo 2: number analyzed (Participants) | 107 | 213 | 107 | 222 | 105 | 218 | 307 | 109
  NZ98/254 Mo 2 | 57 [47 to 67] | 52 [45 to 59] | 89 [81 to 94] | 93 [89 to 96] | 51 [41 to 61] | 57 [50 to 64] | 93 [89 to 95] | 7 [3 to 14]
  NZ98/254 Mo 3: number analyzed (Participants) | 107 | 208 | 104 | 215 | 104 | 215 | 301 | 108
  NZ98/254 Mo 3 | 50 [40 to 59] | 43 [36 to 50] | 78 [69 to 85] | 81 [76 to 86] | 91 [84 to 96] | 91 [86 to 94] | 93 [90 to 96] | 6 [3 to 13]
  NZ98/254 Mo 7: number analyzed (Participants) | 86 | 172 | 94 | 187 | 91 | 179 | 254 | 95
  NZ98/254 Mo 7 | 94 [87 to 98] | 27 [21 to 35] | 95 [88 to 98] | 62 [55 to 69] | 92 [85 to 97] | 69 [62 to 76] | 75 [69 to 80] | 77 [67 to 85]

6. Secondary Outcome: Geometric Mean Titers (GMTs) After Primary and Booster Vaccination.
Description: Immunogenicity was evaluated by measuring the Geometric mean titers (GMTs) after primary and booster vaccination against 44/76-SL, 5/99, NZ98/254.
Time Frame: month-1, month-2, month-3, month-6 and month-7
Population: Analysis was performed as per the protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 334 | 116
Titers
  44/76 GMT Mo 0 | 3.41 [2.54 to 4.58] | 4.24 [3.44 to 5.22] | 3.34 [2.49 to 4.48] | 3.35 [2.72 to 4.11] | 3.39 [2.52 to 4.56] | 3.99 [3.25 to 4.9] | 3.87 [3.26 to 4.6] | 3.89 [2.91 to 5.19]
  44/76 GMT Mo 1: number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  44/76 GMT Mo 1 | 46 [33 to 63] | 58 [46 to 72] | 56 [40 to 77] | 52 [41 to 65] | 44 [32 to 61] | 57 [45 to 71] | 60 [49 to 72] | 3.39 [2.46 to 4.65]
  44/76 GMT Mo 2: number analyzed (Participants) | 108 | 213 | 108 | 222 | 105 | 219 | 307 | 109
  44/76 GMT Mo 2 | 31 [23 to 41] | 41 [34 to 50] | 182 [138 to 240] | 187 [154 to 228] | 28 [21 to 37] | 38 [31 to 46] | 193 [164 to 228] | 4.09 [3.11 to 5.38]
  44/76 GMT Mo 3: number analyzed (Participants) | 107 | 208 | 105 | 215 | 104 | 215 | 303 | 108
  44/76 GMT Mo 3 | 20 [16 to 26] | 31 [26 to 38] | 132 [101 to 172] | 114 [95 to 137] | 182 [139 to 236] | 230 [191 to 277] | 240 [205 to 280] | 4.04 [3.12 to 5.22]
  44/76 GMT Mo 6: number analyzed (Participants) | 100 | 188 | 100 | 198 | 99 | 201 | 278 | 100
  44/76 GMT Mo 6 | 13 [9.24 to 18] | 15 [12 to 19] | 59 [43 to 82] | 50 [39 to 63] | 54 [39 to 75] | 75 [60 to 95] | 86 [70 to 104] | 3.9 [2.82 to 5.4]
  44/76 GMT Mo 7: number analyzed (Participants) | 86 | 173 | 95 | 186 | 91 | 179 | 255 | 95
  44/76 GMT Mo 7 | 218 [157 to 302] | 12 [9.69 to 15] | 324 [236 to 443] | 36 [29 to 45] | 259 [188 to 357] | 48 [38 to 60] | 59 [49 to 72] | 56 [41 to 77]
  5/99 GMT Mo 0 | 2.61 [2.03 to 3.34] | 3.15 [2.64 to 3.75] | 2.59 [2.02 to 3.32] | 2.52 [2.11 to 2.99] | 2.43 [1.89 to 3.12] | 2.72 [2.29 to 3.24] | 2.58 [2.23 to 2.98] | 2.27 [1.78 to 2.89]
  5/99 GMT Mo 1: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  5/99 GMT Mo 1 | 81 [61 to 109] | 64 [52 to 79] | 66 [49 to 88] | 72 [59 to 88] | 57 [42 to 76] | 76 [62 to 93] | 71 [60 to 84] | 2.56 [1.93 to 3.4]
  5/99 GMT Mo 2: number analyzed (Participants) | 108 | 213 | 108 | 222 | 105 | 219 | 308 | 109
  5/99 GMT Mo 2 | 40 [31 to 51] | 34 [28 to 40] | 505 [396 to 644] | 451 [381 to 535] | 26 [20 to 33] | 40 [34 to 48] | 481 [415 to 556] | 2.48 [1.95 to 3.16]
  5/99 GMT Mo 3: number analyzed (Participants) | 107 | 209 | 105 | 215 | 105 | 215 | 303 | 108
  5/99 GMT Mo 3 | 25 [20 to 31] | 23 [20 to 27] | 303 [242 to 380] | 273 [233 to 320] | 540 [431 to 677] | 822 [702 to 964] | 584 [510 to 668] | 2.58 [2.07 to 3.22]
  5/99 GMT Mo 6: number analyzed (Participants) | 100 | 188 | 100 | 198 | 99 | 201 | 278 | 100
  5/99 GMT Mo 6 | 12 [9.56 to 16] | 11 [9.26 to 13] | 125 [98 to 160] | 113 [95 to 135] | 124 [97 to 158] | 147 [123 to 175] | 186 [160 to 216] | 2.03 [1.59 to 2.59]
  5/99 GMT Mo 7: number analyzed (Participants) | 86 | 173 | 95 | 187 | 91 | 179 | 255 | 95
  5/99 GMT Mo 7 | 880 [675 to 1147] | 8.61 [7.13 to 10] | 1094 [849 to 1410] | 99 [82 to 119] | 994 [767 to 1289] | 121 [101 to 146] | 164 [141 to 192] | 53 [41 to 68]
  NZ98/254 GMT Mo 0: number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 333 | 116
  NZ98/254 GMT Mo 0 | 2.87 [2.14 to 3.84] | 3.35 [2.72 to 4.13] | 3.43 [2.56 to 4.59] | 2.98 [2.43 to 3.66] | 3.07 [2.28 to 4.12] | 3.39 [2.76 to 4.16] | 2.83 [2.38 to 3.36] | 3.12 [2.34 to 4.15]
  NZ98/254 GMT Mo1: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  NZ98/254 GMT Mo1 | 42 [31 to 56] | 44 [36 to 55] | 47 [35 to 63] | 45 [36 to 55] | 37 [27 to 50] | 42 [34 to 52] | 49 [41 to 58] | 2.85 [2.11 to 3.84]
  NZ98/254 GMT Mo 2: number analyzed (Participants) | 107 | 213 | 108 | 222 | 105 | 218 | 308 | 109
  NZ98/254 GMT Mo 2 | 23 [17 to 30] | 25 [20 to 31] | 98 [72 to 132] | 89 [72 to 110] | 19 [14 to 26] | 26 [21 to 32] | 92 [77 to 110] | 3.28 [2.43 to 4.41]
  NZ98/254 GMT Mo 3: number analyzed (Participants) | 107 | 208 | 105 | 215 | 104 | 215 | 302 | 108
  NZ98/254 GMT Mo 3 | 17 [13 to 22] | 19 [16 to 24] | 61 [46 to 82] | 52 [42 to 64] | 117 [87 to 157] | 125 [102 to 154] | 122 [102 to 145] | 3.57 [2.68 to 4.75]
  NZ98/254 GMT Mo 6: number analyzed (Participants) | 99 | 188 | 100 | 198 | 99 | 200 | 278 | 100
  NZ98/254 GMT Mo 6 | 12 [8.94 to 17] | 11 [8.63 to 14] | 31 [22 to 42] | 29 [23 to 36] | 44 [32 to 61] | 49 [39 to 61] | 52 [43 to 63] | 4.17 [3.04 to 5.72]
  NZ98/254 GMT Mo 7: number analyzed (Participants) | 86 | 172 | 95 | 187 | 91 | 179 | 255 | 95
  NZ98/254 GMT Mo 7 | 140 [101 to 195] | 10 [8.01 to 13] | 181 [132 to 248] | 24 [19 to 30] | 168 [122 to 232] | 39 [31 to 49] | 41 [34 to 50] | 47 [34 to 64]

7. Secondary Outcome: Geometric Mean Ratios (GMRs) After Primary and Booster Vaccination.
Description: Immunogenicity was evaluated by measuring the Geometric mean ratios (GMRs) after primary and booster vaccination against 44/76-SL, 5/99, NZ98/254.
Time Frame: month-1, month-2, month-3, month-6 and month-7
Population: Analysis was performed as per the protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 112 | 223 | 113 | 231 | 110 | 232 | 333 | 115
Ratio
  44/76 GMR Mo 1 to 0 | 13 [10 to 18] | 14 [11 to 17] | 17 [12 to 22] | 16 [13 to 19] | 13 [9.71 to 18] | 14 [12 to 17] | 15 [13 to 18] | 0.89 [0.66 to 1.18]
  44/76 GMR Mo 2 to 0: number analyzed (Participants) | 108 | 213 | 107 | 222 | 105 | 219 | 307 | 109
  44/76 GMR Mo 2 to 0 | 8.92 [6.73 to 12] | 9.65 [7.88 to 12] | 53 [40 to 71] | 56 [46 to 69] | 8.43 [6.33 to 11] | 9.51 [7.79 to 12] | 50 [42 to 59] | 1.04 [0.79 to 1.38]
  44/76 GMR Mo 3 to 0: number analyzed (Participants) | 107 | 208 | 104 | 215 | 104 | 215 | 303 | 108
  44/76 GMR Mo 3 to 0 | 5.98 [4.51 to 7.92] | 7.31 [5.97 to 8.96] | 37 [28 to 50] | 34 [28 to 42] | 55 [41 to 73] | 58 [48 to 71] | 62 [52 to 73] | 0.98 [0.74 to 1.3]
  44/76 GMR Mo 6 to 0: number analyzed (Participants) | 100 | 188 | 99 | 198 | 99 | 201 | 278 | 100
  44/76 GMR Mo 6 to 0 | 3.98 [2.96 to 5.35] | 3.64 [2.93 to 4.52] | 17 [13 to 23] | 16 [13 to 19] | 16 [12 to 21] | 20 [16 to 25] | 23 [19 to 27] | 0.92 [0.69 to 1.24]
  44/76 GMR Mo 7 to 0: number analyzed (Participants) | 86 | 173 | 94 | 186 | 91 | 179 | 255 | 95
  44/76 GMR Mo 7 to 0 | 74 [54 to 103] | 3.09 [2.46 to 3.88] | 92 [67 to 125] | 12 [9.24 to 14] | 79 [58 to 109] | 13 [11 to 17] | 16 [13 to 19] | 13 [9.76 to 18]
  44/76 GMR Mo 7 to 6: number analyzed (Participants) | 86 | 173 | 95 | 186 | 91 | 179 | 255 | 94
  44/76 GMR Mo 7 to 6 | 18 [14 to 23] | 0.89 [0.76 to 1.05] | 5.36 [4.3 to 6.68] | 0.72 [0.61 to 0.84] | 5.08 [4.05 to 6.37] | 0.67 [0.57 to 0.79] | 0.67 [0.59 to 0.77] | 14 [11 to 17]
  5/99 GMR Mo 1 to 0: number analyzed (Participants) | 111 | 223 | 113 | 231 | 110 | 232 | 333 | 115
  5/99 GMR Mo 1 to 0 | 31 [23 to 42] | 20 [16 to 25] | 25 [19 to 34] | 29 [23 to 35] | 23 [17 to 32] | 28 [23 to 34] | 28 [23 to 33] | 1.13 [0.84 to 1.52]
  5/99 GMR Mo 2 to 0: number analyzed (Participants) | 108 | 213 | 107 | 222 | 105 | 219 | 308 | 109
  5/99 GMR Mo 2 to 0 | 15 [11 to 20] | 11 [8.65 to 13] | 198 [149 to 262] | 181 [149 to 220] | 11 [8.13 to 14] | 15 [12 to 18] | 186 [158 to 220] | 1.06 [0.8 to 1.4]
  5/99 GMR Mo 3 to 0: number analyzed (Participants) | 107 | 209 | 104 | 215 | 105 | 215 | 303 | 108
  5/99 GMR Mo 3 to 0 | 9.22 [6.94 to 12] | 7.37 [6.01 to 9.04] | 115 [86 to 153] | 109 [89 to 133] | 233 [175 to 311] | 306 [250 to 374] | 225 [190 to 267] | 1.09 [0.82 to 1.44]
  5/99 GMR Mo 6 to 0: number analyzed (Participants) | 100 | 188 | 99 | 198 | 99 | 201 | 278 | 100
  5/99 GMR Mo 6 to 0 | 4.65 [3.47 to 6.23] | 3.83 [3.09 to 4.75] | 49 [37 to 66] | 45 [36 to 55] | 52 [39 to 70] | 56 [45 to 69] | 74 [62 to 88] | 0.82 [0.61 to 1.1]
  5/99 GMR Mo 7 to 0: number analyzed (Participants) | 86 | 173 | 94 | 187 | 91 | 179 | 255 | 95
  5/99 GMR Mo 7 to 0 | 355 [254 to 497] | 3.07 [2.42 to 3.89] | 430 [312 to 594] | 40 [32 to 50] | 427 [307 to 593] | 46 [36 to 58] | 65 [53 to 79] | 21 [16 to 29]
  5/99 GMR Mo 7 to 6: number analyzed (Participants) | 86 | 173 | 95 | 187 | 91 | 179 | 255 | 94
  5/99 GMR Mo 7 to 6 | 71 [55 to 90] | 0.83 [0.7 to 0.99] | 8.98 [7.13 to 11] | 0.87 [0.74 to 1.03] | 7.92 [6.26 to 10] | 0.83 [0.71 to 0.99] | 0.86 [0.74 to 0.99] | 26 [20 to 32]
  NZ98/254 GMR Mo 1 to 0 | 14 [11 to 19] | 13 [11 to 16] | 14 [10 to 18] | 15 [12 to 18] | 12 [9 to 16] | 12 [10 to 15] | 17 [15 to 21] | 0.91 [0.68 to 1.2]
  NZ98/254 GMR Mo 2 to 0 | 7.69 [5.86 to 10] | 7.24 [5.97 to 8.79] | 29 [22 to 38] | 30 [24 to 36] | 6.46 [4.91 to 8.5] | 7.96 [6.57 to 9.63] | 33 [28 to 39] | 1.06 [0.81 to 1.38]
  NZ98/254 GMR Mo 3 to 0 | 6.01 [4.54 to 7.96] | 5.5 [4.49 to 6.74] | 18 [14 to 24] | 18 [14 to 21] | 40 [30 to 54] | 38 [32 to 47] | 44 [37 to 52] | 1.13 [0.86 to 1.5]
  NZ98/254 GMR Mo 6 to 0: number analyzed (Participants) | 99 | 188 | 99 | 198 | 99 | 200 | 277 | 100
  NZ98/254 GMR Mo 6 to 0 | 4.75 [3.62 to 6.24] | 3.49 [2.86 to 4.26] | 9.26 [7.05 to 12] | 10 [8.29 to 12] | 14 [11 to 19] | 15 [13 to 19] | 19 [16 to 22] | 1.28 [0.98 to 1.68]
  NZ98/254 GMR Mo 7 to 0: number analyzed (Participants) | 86 | 172 | 94 | 187 | 91 | 179 | 254 | 95
  NZ98/254 GMR Mo 7 to 0 | 59 [44 to 80] | 3.32 [2.67 to 4.12] | 53 [40 to 71] | 8.94 [7.26 to 11] | 57 [42 to 77] | 13 [10 to 16] | 15 [12 to 18] | 15 [11 to 19]
  NZ98/254 GMR Mo 7 to 6: number analyzed (Participants) | 85 | 172 | 95 | 187 | 91 | 179 | 255 | 94
  NZ98/254 GMR Mo 7 to 6 | 11 [8.73 to 14] | 0.99 [0.84 to 1.17] | 5.86 [4.7 to 7.3] | 0.85 [0.73 to 1] | 3.95 [3.15 to 4.95] | 0.84 [0.72 to 0.99] | 0.81 [0.7 to 0.92] | 11 [8.98 to 14]

8. Secondary Outcome: GMCs of Antibodies Against 287-953Antigen (ELISA) After Primary and Booster Vaccination.
Description: Immunogenicity was evaluated by measuring the Geometric mean Concentration (GMCs) after primary and booster vaccination against Antigen 287-953 Antigen.
Time Frame: month-1, month-2, month-3, month-6 and month-7
Population: Analysis was performed as per the protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 34 | 35 | 35 | 35 | 35 | 35 | 35 | 35
IU/ml
  GMC Mo 0: number analyzed (Participants) | 34 | 35 | 35 | 32 | 35 | 35 | 35 | 35
  GMC Mo 0 | 35 [25 to 51] | 35 [25 to 50] | 43 [30 to 61] | 37 [26 to 54] | 44 [31 to 63] | 32 [23 to 46] | 32 [22 to 45] | 48 [34 to 68]
  GMC Mo 1 | 190 [113 to 318] | 204 [123 to 340] | 334 [200 to 555] | 217 [130 to 361] | 234 [140 to 389] | 220 [132 to 367] | 521 [313 to 868] | 50 [30 to 82]
  GMC Mo 2: number analyzed (Participants) | 34 | 35 | 35 | 34 | 35 | 35 | 35 | 35
  GMC Mo 2 | 173 [115 to 261] | 154 [102 to 231] | 3025 [2015 to 4543] | 3875 [2566 to 5854] | 175 [117 to 263] | 144 [96 to 216] | 3693 [2459 to 5545] | 42 [28 to 62]
  GMC Mo 3: number analyzed (Participants) | 34 | 35 | 35 | 34 | 35 | 35 | 35 | 35
  GMC Mo 3 | 102 [69 to 152] | 124 [84 to 183] | 1612 [1093 to 2378] | 1831 [1234 to 2716] | 3332 [2259 to 4916] | 2936 [1990 to 4332] | 5314 [3602 to 7839] | 42 [29 to 62]
  GMC Mo 6 | 91 [59 to 138] | 72 [48 to 110] | 565 [372 to 857] | 488 [322 to 741] | 807 [531 to 1224] | 628 [414 to 953] | 1602 [1055 to 2431] | 37 [24 to 56]
  GMC Mo 7: number analyzed (Participants) | 34 | 34 | 35 | 34 | 35 | 35 | 35 | 35
  GMC Mo 7 | 2240 [1385 to 3623] | 69 [43 to 112] | 3840 [2391 to 6168] | 383 [237 to 620] | 5492 [3419 to 8821] | 532 [331 to 855] | 1111 [692 to 1785] | 283 [176 to 454]

9. Secondary Outcome: GMRs of Antibodies Against 287-953Antigen (ELISA) After Primary and Booster Vaccination
Description: Immunogenicity was evaluated by measuring the Geometric mean Ratios (GMRs) after primary and booster vaccination against 287-953Antigen
Time Frame: month-1, month-2, month-3, month-6 and month-7
Population: Analysis was performed as per the protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 34 | 35 | 35 | 35 | 35 | 35 | 35 | 35
Ratio
  GMR Mo 1 to 0: number analyzed (Participants) | 34 | 35 | 35 | 32 | 35 | 35 | 35 | 35
  GMR Mo 1 to 0 | 5.73 [3.19 to 9.05] | 5.82 [3.48 to 9.73] | 7.75 [4.64 to 13] | 5.34 [3.12 to 9.14] | 5.26 [3.14 to 8.79] | 6.85 [4.09 to 11] | 16 [9.77 to 27] | 1.03 [0.62 to 1.73]
  GMR Mo 2 to 0: number analyzed (Participants) | 34 | 35 | 35 | 31 | 35 | 35 | 35 | 35
  GMR Mo 2 to 0 | 4.9 [3.2 to 7.5] | 4.38 [2.88 to 6.66] | 70 [46 to 107] | 112 [72 to 175] | 3.94 [2.59 to 5.99] | 4.46 [2.93 to 6.79] | 116 [76 to 176] | 0.87 [0.57 to 1.32]
  GMR Mo 3 to 0: number analyzed (Participants) | 34 | 35 | 35 | 31 | 35 | 35 | 35 | 35
  GMR Mo 3 to 0 | 2.9 [1.82 to 4.61] | 3.54 [2.24 to 5.59] | 37 [24 to 59] | 55 [34 to 89] | 75 [47 to 118] | 91 [58 to 144] | 167 [105 to 263] | 0.88 [0.56 to 1.4]
  GMR Mo 6 to 0: number analyzed (Participants) | 34 | 35 | 35 | 32 | 35 | 35 | 35 | 35
  GMR Mo 6 to 0 | 2.56 [1.59 to 4.13] | 2.06 [1.29 to 3.3] | 13 [8.2 to 21] | 13 [7.86 to 21] | 18 [11 to 29] | 20 [12 to 31] | 50 [31 to 80] | 0.77 [0.48 to 1.23]
  GMR Mo 7 to 0: number analyzed (Participants) | 34 | 34 | 35 | 31 | 35 | 35 | 35 | 35
  GMR Mo 7 to 0 | 63 [34 to 119] | 1.94 [1.03 to 3.64] | 89 [48 to 166] | 11 [5.67 to 21] | 123 [66 to 229] | 17 [8.9 to 31] | 35 [19 to 65] | 5.9 [3.17 to 11]

10. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs Throughout the Study.
Description: Safety was assessed as the number of subjects who reported unsolicited AEs throughout the study.
Time Frame: Throughout the study
Population: Analysis was performed as per the safety dataset.
Measure: Number; unit: participants
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 128 | 247 | 128 | 247 | 127 | 253 | 373 | 128
participants
  Any AE's | 65 | 137 | 73 | 143 | 72 | 148 | 210 | 80
  At least possibly related AEs | 22 | 36 | 30 | 36 | 24 | 43 | 76 | 26
  Serious AEs | 5 | 4 | 2 | 4 | 2 | 4 | 11 | 3
  At least possibly related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  AEs leading to discontinuation | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0

11. Post Hoc Outcome: Percentage of Subjects With hSBA Titers≥4 After Receiving Second Dose of Vaccination
Description: Immunogenicity was evaluated by measuring the percentage of subjects with hSBA titter >1:4 against M10713 strain at 1 month after second dose of vaccination (Month 3)
Time Frame: At one month after second dose (Month 3)
Population: Analysis was performed as per the protocol dataset. Only groups rMenB01 and rMenB02 are applicable to this endpoint as the post-hoc outcome was assessed at an interval of 1 month (rMenB01) or 2 months (rMenB02 ) to kill M10713 strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB01 | rMenB02
Number analyzed (Participants) | 46 | 46
Percentage of subjects
  Baseline | 96 [85 to 99] | 80 [66 to 91]
  1 month after second dose | 100 [92 to 100] | 100 [92 to 100]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were collected from Day 1 through 7,Serious AEs were collected throughout the study.
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Serious Adverse Events (participants affected / at risk) | 5/128 | 4/247 | 2/128 | 4/247 | 2/127 | 4/253 | 11/373 | 3/128
Other Adverse Events (participants affected / at risk) | 123/128 | 238/247 | 126/128 | 242/247 | 118/127 | 240/253 | 354/373 | 125/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rMenB06 (N=128) | rMenB0 (N=247) | rMenB016 (N=128) | rMenB01 (N=247) | rMenB026 (N=127) | rMenB02 (N=253) | rMenB012 (N=373) | rMenB6 (N=128)
APPENDICITIS (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1
DYSENTERY (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MENINGITIS BACTERlAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PNEUMONIA VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SHIGELLAIN FECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOXICITY TO VARlOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
JUVENILE IDIOPATHIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
ADENOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BENGIN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CONVULSION (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
EPILEPSY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PREMATURE LABOUR (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PANIC ATTACK (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
GLOMERULONEPHRITIS MINIMAL LESION (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TESTICULAR TORSION (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ADENOIDECTOMY (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TONSILLECTOMY (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB06 (N=128) | rMenB0 (N=247) | rMenB016 (N=128) | rMenB01 (N=247) | rMenB026 (N=127) | rMenB02 (N=253) | rMenB012 (N=373) | rMenB6 (N=128)
NAUSEA (Gastrointestinal disorders) | 41 (80) | 80 (120) | 51 (109) | 72 (126) | 42 (72) | 89 (156) | 143 (276) | 49 (90)
INJECTION SITE ERYTHEMA (General disorders) | 93 (211) | 162 (338) | 97 (225) | 188 (428) | 94 (251) | 172 (389) | 282 (680) | 86 (169)
INJECTION SITE INDURATION (General disorders) | 72 (149) | 130 (240) | 76 (167) | 151 (328) | 82 (191) | 122 (234) | 228 (564) | 58 (116)
INJECTION SITE PAIN (General disorders) | 122 (378) | 236 (667) | 124 (396) | 237 (729) | 113 (398) | 236 (749) | 345 (1160) | 123 (398)
INJECTION SITE SWELLING (General disorders) | 73 (129) | 132 (244) | 81 (172) | 144 (310) | 76 (171) | 115 (242) | 226 (523) | 55 (92)
MALAISE (General disorders) | 92 (222) | 181 (371) | 96 (238) | 172 (405) | 87 (235) | 185 (444) | 272 (690) | 89 (205)
PYREXIA (General disorders) | 12 (17) | 8 (11) | 13 (18) | 21 (22) | 18 (20) | 26 (30) | 38 (50) | 20 (27)
BRONCHITIS (Infections and infestations) | 6 (6) | 7 (7) | 5 (5) | 10 (10) | 9 (9) | 6 (6) | 14 (14) | 11 (14)
GASTROENTERITIS (Infections and infestations) | 4 (4) | 7 (8) | 2 (2) | 15 (15) | 2 (2) | 14 (15) | 23 (27) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 9 (9) | 24 (26) | 18 (18) | 20 (21) | 9 (11) | 28 (30) | 43 (46) | 13 (15)
PHARYNGITIS (Infections and infestations) | 7 (7) | 11 (11) | 5 (6) | 9 (10) | 4 (4) | 7 (7) | 21 (24) | 8 (9)
TONSILLITIS (Infections and infestations) | 3 (4) | 5 (5) | 4 (5) | 7 (9) | 3 (3) | 6 (7) | 16 (18) | 7 (8)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 4 (4) | 6 (6) | 3 (3) | 7 (8) | 7 (7) | 7 (7) | 15 (15) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 56 (101) | 76 (131) | 55 (106) | 81 (175) | 39 (81) | 105 (215) | 146 (320) | 44 (77)
MYALGIA (Musculoskeletal and connective tissue disorders) | 85 (170) | 141 (266) | 91 (187) | 158 (335) | 82 (193) | 160 (357) | 238 (568) | 91 (198)
HEADACHE (Nervous system disorders) | 79 (185) | 140 (346) | 88 (256) | 160 (444) | 74 (208) | 165 (452) | 244 (704) | 76 (209)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.